CLINICAL TRIAL: NCT01352637
Title: Enhancing Exposure Therapy for PTSD: Virtual Reality and Imaginal Exposure With a Cognitive Enhancer
Brief Title: Enhancing Exposure Therapy for Post Traumatic Stress Disorder (PTSD): Virtual Reality and Imaginal Exposure With a Cognitive Enhancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Emory University (Other); University of Southern California (Other); VA Long Beach Healthcare System (U.S. Federal Agency); National Intrepid Center of Excellence (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1005011047
Record Dates: First submitted 2011-02-18; First posted 2011-05-12 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Traumatic Event; Trauma Survivor; Exposure Therapy; PTSD DCS; Virtual Reality Exposure; Veteran; Combat-related PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cycloserine

STUDY DESIGN:
Intervention Model Description: The two primary co-aims of this study are
  1. to examine the effects of DCS versus placebo (PLA) augmentation of exposure therapy on PTSD symptoms and
  2. to examine the relative efficacy of virtual reality enhanced exposure therapy (VRE) and exposure therapy (PE) on PTSD symptoms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo + Prolonged Imaginal Exposure (Placebo Comparator): Drug: Placebo (sugar pill) + Prolonged Imaginal Exposure (PE) PTSD treatment
  Interventions: Drug: Placebo + Prolonged Imaginal Exposure
- Placebo + VR exposure (Placebo Comparator): Drug: Placebo (sugar pill) + Virtual Reality Exposure (VR) PTSD treatment
  Interventions: Drug: Placebo (sugar pill) + Virtual Reality Exposure
- DCS + Prolonged Imaginal Exposure (Active Comparator): Drug: 50mg DCS (D-Cycloserine ) + Prolonged Imaginal Exposure (PE) PTSD treatment
  Interventions: Drug: DCS (D-Cycloserine ) + Prolonged Imaginal Exposure
- DCS+VR exposure (Active Comparator): Drug: 50mg DCS (D-Cycloserine ) + Virtual Reality Exposure (VR) PTSD treatment
  Interventions: Drug: DCS (D-Cycloserine ) + Virtual Reality Exposure

INTERVENTIONS:
Drug: DCS (D-Cycloserine ) + Prolonged Imaginal Exposure — 50mg DCS (taken once a week on the day of the therapy session) + Prolonged Imaginal Exposure
  Arms: DCS + Prolonged Imaginal Exposure
Drug: DCS (D-Cycloserine ) + Virtual Reality Exposure — 50mg DCS (taken once a week on the day of the therapy session) + Virtual Reality Exposure
  Arms: DCS+VR exposure
Drug: Placebo + Prolonged Imaginal Exposure — Placebo (taken once a week on the day of the therapy session) + Prolonged Imaginal Exposure
  Arms: Placebo + Prolonged Imaginal Exposure
Drug: Placebo (sugar pill) + Virtual Reality Exposure — Placebo (taken once a week on the day of the therapy session) + Virtual Reality Exposure
  Arms: Placebo + VR exposure

SUMMARY:
The purpose of this study is to test the differences between four active treatment conditions for combat-related Post Traumatic Stress Disorder (PTSD): virtual reality exposure therapy (VRE) or prolonged imaginal exposure therapy (PE), both with DCS or placebo, as well as to examine predictors for PTSD and response to treatment in active duty military personnel, veterans, and civilians who served in Iraq and Afghanistan.

DETAILED DESCRIPTION:
Post Traumatic Stress Disorder (PTSD) is an anxiety disorder that can develop following exposure to traumatic events and includes symptoms of re-experiencing the trauma, such as through nightmares and flashbacks, avoidance and numbing, and physical hyperarousal. PTSD has been estimated to affect 10-20% of returning Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) veterans. The most effective intervention found for PTSD is exposure therapy, which can be delivered in different formats, e. g. via virtual reality (VR) and as imaginal exposure. The goal of this study is to test the difference between 4 study conditions: virtual reality exposure therapy (VRE) or prolonged imaginal exposure therapy (PE), both combined with an antibiotic drug, DCS (active pill vs. placebo). D-Cycloserine (DCS), a drug that has been FDA approved for over 20 years, has been hypothesized to enhance the therapeutic effects of exposure therapy.). A secondary purpose of this study is to examine predictors for PTSD and response to PTSD intervention in active duty military personnel, veterans, and civilians who served in Iraq/Afghanistan. Psychophysiological factors (e.g. heart rate, blood pressure) and/or a genetic polymorphism (BDNF Val66Met) obtained from a saliva sample will be examined.

The two primary co-aims are

1. to examine the effects of DCS versus placebo (PLA) augmentation of exposure therapy on PTSD symptoms, and
2. to examine the relative efficacy of virtual reality enhanced exposure therapy (VRE) and exposure therapy (PE) on PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OEF-OIF (Operations Enduring Freedom or Iraqi Freedom) Combat Related PTSD;
2. Female participants of childbearing potential must agree to use an effective method of birth control (i.e., oral contraceptive, Norplant, diaphragm, condom, or spermicide) during the course of the study, or to remain abstinent from sex, to ensure they do not become pregnant during the course of the study;
3. Ability to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments;
4. Participants must be literate in English;
5. Patients must be medically healthy and willing to take the study drug;
6. VRE stimuli available must be consistent with subject's trauma.

Exclusion Criteria:

1. Lifetime or current diagnosis of schizophrenia or other psychotic disorder, bipolar disorder;
2. Participation in a clinical trial during the previous 3 months;
3. Current evidence or history of significant unstable medical illness or organic brain impairment, including stroke, CNS tumor, demyelinating disease, cardiac, pulmonary, gastrointestinal, renal or hepatic impairment;
4. Patients who in the investigator's judgment pose a current suicidal or homicidal risk;
5. Alcohol, medication, or illegal substance dependence within the past 90 days;
6. Treatment with any other concomitant medication with primarily CNS activity, or treatment with any medication that the PI judges not acceptable for this study;
7. history of seizures;
8. Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, Ph.D., Principal Investigator — Weill Medical College of Cornell University; Barbara Rothbaum, Ph.D., ABPP, Principal Investigator — Emory University; Skip Rizzo, Ph. D., Principal Investigator — University of Southern California
Locations (5):
- United States (5):
  - VA Long Beach Healthcare System, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Walter Reed Army Medical Center/National Intrepid Center of Excellence (NICoE), Bethesda, Maryland
  - Weill Cornell Medical College, New York, New York

REFERENCES:
- [Derived] Difede J, Rothbaum BO, Rizzo AA, Wyka K, Spielman L, Reist C, Roy MJ, Jovanovic T, Norrholm SD, Cukor J, Olden M, Glatt CE, Lee FS. Enhancing exposure therapy for posttraumatic stress disorder (PTSD): a randomized clinical trial of virtual reality and imaginal exposure with a cognitive enhancer. Transl Psychiatry. 2022 Jul 27;12(1):299. doi: 10.1038/s41398-022-02066-x. PMID 35896533
- [Derived] Difede J, Rothbaum BO, Rizzo AA, Wyka K, Spielman L, Jovanovic T, Reist C, Roy MJ, Norrholm SD, Glatt C, Lee F. Enhanced exposure therapy for combat-related Posttraumatic Stress Disorder (PTSD): Study protocol for a randomized controlled trial. Contemp Clin Trials. 2019 Dec;87:105857. doi: 10.1016/j.cct.2019.105857. Epub 2019 Oct 24. PMID 31669451
- See also: Related Info — http://www.patss.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total sample size is n=192. Randomization allocation ratio was 1:1:1:1 to VRE vs. PE and DCS vs. placebo.
  Study had 2 co-primary aims to examine:
  1. the effects of DCS (n=95) vs placebo (n=97) augmentation of exposure therapy
  2. the relative efficacy of VRE (n=97) and PE (n=95) on PTSD symptoms.
Groups:
- Virtual Reality Exposure (VRE): Virtual Reality Exposure (VRE): PTSD treatment
- Prolonged Imaginal Exposure (PE): Drug: Placebo (sugar pill) + Virtual Reality Exposure (VR) PTSD treatment
  Prolonged Imaginal Exposure (PE): PTSD treatment
- Drug: D-Cycloserine (DCS): D-Cycloserine (DCS) (taken once a week on the day of the therapy session)
- Drug: Placebo: Drug: Placebo (sugar pill) (taken once a week on the day of the therapy session)
Period: Exposure Therapy
Arm/Group | Virtual Reality Exposure (VRE) | Prolonged Imaginal Exposure (PE) | Drug: D-Cycloserine (DCS) | Drug: Placebo
Started | 97 | 95 | 0 | 0
Completed | 70 | 62 | 0 | 0
Not Completed | 27 | 33 | 0 | 0
Period: Drug
Arm/Group | Virtual Reality Exposure (VRE) | Prolonged Imaginal Exposure (PE) | Drug: D-Cycloserine (DCS) | Drug: Placebo
Started | 0 | 0 | 95 | 97
Completed | 0 | 0 | 70 | 62
Not Completed | 0 | 0 | 25 | 35

BASELINE CHARACTERISTICS:
Population: Total sample size is n=192. Randomization allocation ratio was 1:1:1:1 to VRE vs. PE and DCS vs. placebo.
  Study had 2 co-primary aims to examine:
  1. the effects of DCS (n=95) vs placebo (n=97) augmentation of exposure therapy
  2. the relative efficacy of VRE (n=97) and PE (n=95) on PTSD symptoms.
Groups:
- Virtual Reality Exposure (VRE)+Drug: DCycloserine (DCS): Virtual Reality Exposure (VRE): PTSD treatment + D-Cycloserine (DCS) (taken once a week on the day of the therapy session)
- Prolonged Imaginal Exposure (PE)+Drug: DCycloserine (DCS): Prolonged Imaginal Exposure (PE): PTSD treatment + D-Cycloserine (DCS) (taken once a week on the day of the therapy session)
- Virtual Reality Exposure (VRE)+Drug: Placebo: Virtual Reality Exposure (VRE): PTSD treatment + Placebo (sugar pill) (taken once a week on the day of the therapy session)
- Prolonged Imaginal Exposure (PE)+Drug: Placebo: Prolonged Imaginal Exposure (PE): PTSD treatment + Placebo (sugar pill) (taken once a week on the day of the therapy session)
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Exposure (VRE)+Drug: DCycloserine (DCS) | Prolonged Imaginal Exposure (PE)+Drug: DCycloserine (DCS) | Virtual Reality Exposure (VRE)+Drug: Placebo | Prolonged Imaginal Exposure (PE)+Drug: Placebo | Total
Number analyzed (Participants) | 47 | 48 | 50 | 47 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.74 (7.69) | 36.17 (8.53) | 34.80 (6.99) | 33.70 (7.95) | 34.62 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 5 | 20
  Male | 41 | 42 | 47 | 42 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 21 | 26 | 21 | 88
  African American/Black | 8 | 6 | 6 | 9 | 29
  Hispanic/Latino | 16 | 14 | 10 | 13 | 53
  Other | 3 | 7 | 8 | 4 | 22
CAPS-IV, past week [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale (CAPS) for the DSM-IV [34]. The CAPS-IV is a structured clinical interview designed to assess the 17 DSM-IV PTSD symptoms. CAPS-IV provides categorical ratings of diagnostic status as well as a quantitative index of symptom severity. The CAPS total severity score is based on response to the 17 items that assess the frequency and intensity of current PTSD symptoms. Symptom severity is assessed separately for past month and past week time frames.
  CAPS-IV range is 0-136, higher scores mean a worse outcome.
  units on a scale | 71.72 (19.98) | 75.08 (18.69) | 74.46 (19.11) | 70.74 (200.37) | 73.04 (19.47)

OUTCOME MEASURES:

1. Primary Outcome: CAPS-IV at the End of Treatment
Description: Clinician Administered PTSD Scale (CAPS) for the DSM-IV [34]. The CAPS-IV is a structured clinical interview designed to assess the 17 DSM-IV PTSD symptoms. CAPS-IV provides categorical ratings of diagnostic status as well as a quantitative index of symptom severity. The CAPS total severity score is based on response to the 17 items that assess the frequency and intensity of current PTSD symptoms. Symptom severity is assessed separately for past month and past week time frames.
  CAPS-IV range is 0-136, higher scores mean a worse outcome.
Time Frame: after weekly treatment session 9 (at posttreatment assessment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prolonged Imaginal Exposure (PE): Prolonged Imaginal Exposure (PE): PTSD treatment
Arm/Group | Virtual Reality Exposure (VRE) | Prolonged Imaginal Exposure (PE) | Drug: D-Cycloserine (DCS) | Drug: Placebo
Number analyzed (Participants) | 97 | 95 | 95 | 97
units on a scale | 52.42 (26.55) | 50.61 (25.22) | 54.20 (26.72) | 48.59 (24.71)

ADVERSE EVENTS:
Time Frame: During treatment (9 weekly therapy sessions).
Description: 18-item Side Effect Screening Checklist was administered at each therapy session to identify possible medication-related side effects and specific adverse symptoms.
Arm/Group | Virtual Reality Exposure (VRE) | Prolonged Imaginal Exposure (PE) | Drug: D-Cycloserine (DCS) | Drug: Placebo
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/95 | 0/95 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/97 | 3/95 | 0/95 | 1/97
Other Adverse Events (participants affected / at risk) | 0/97 | 0/95 | 0/95 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality Exposure (VRE) (N=97) | Prolonged Imaginal Exposure (PE) (N=95) | Drug: D-Cycloserine (DCS) (N=95) | Drug: Placebo (N=97)
Hospitalization (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Cellulitis of the lower extremity
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Chest pains and shortness of breath
Hopitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Injuries due to car accident

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT01352637/Prot_SAP_000.pdf